CLINICAL TRIAL: NCT03943160
Title: Radial accEss for nAvigation to Your CHosen Lesion for Peripheral Vascular Intervention: REACH PVI
Acronym: REACH PVI
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0012-P
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Diamondback 360 Extended Length Orbital Atherectomy System — All patients undergoing peripheral vascular intervention (PVI) via transradial access (TRA) and for whom TRA has been successfully achieved and peripheral lesion deemed appropriate for treatment via TRA per physician discretion.
  Other Names: Stealth 360 Extended Length Orbital Atherectomy System

SUMMARY:
The objective of this study is to evaluate acute clinical results of orbital atherectomy (OA) via radial artery access, including complication rates and cost effectiveness.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively evaluate acute clinical outcomes of orbital atherectomy (OA) via transradial access (TRA) for treatment of peripheral artery disease (PAD) in lower extremity lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years
2. Subject is willing and able to sign the IRB-approved informed consent form (ICF)
3. Subject presents with a Rutherford Classification of 2 to 5
4. Subject has a positive Allen's Test
5. Subject to undergo peripheral angiography and/or PVI via TRA approach per physician discretion

Index Procedure Inclusion Criteria:

1. Physician obtains successful radial artery access (Note: snuffbox access is allowed)
2. Target lesion appropriate (i.e. location/morphology) for OA treatment via TRA within target area
3. OAS use attempted (defined as ViperWire introduced into the body)

Exclusion Criteria:

1. Subject has no palpable radial artery on the planned access arm
2. Subject has a previous failed radial access attempt on planned access arm
3. Subject has a dialysis fistula on planned access arm
4. Subject has a known subclavian stenosis or occlusion
5. Subject has a previous subclavian stent or previous subclavian intervention
6. Subject has a shunt in the radial artery on the planned access arm
7. Subject has evidence of osteomyelitis
8. Subject is currently participating in an investigational drug or device study
9. Subject is pregnant within the study period

Index Procedure Exclusion Criteria

1. Physician unable to obtain radial artery access
2. Physician determines TRA is not acceptable due to patient anatomy, lesion characteristics, and/or disease severity
3. OAS use not attempted (defined as ViperWire introduced into the body)

   Prior to insertion of ViperWire:
4. Femoral access is obtained
5. Unsuccessful peripheral intervention
6. A reportable adverse event has occurred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing peripheral vascular intervention (PVI) via transradial access (TRA) and for whom TRA has been successfully achieved and peripheral lesion deemed appropriate for treatment via TRA per physician discretion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cardiovascular Institute of the South - Lafayette General South West OBL, Lafayette, Louisiana
  - Mercy Hospital, Springfield, Chesterfield, Missouri
  - Columbia University Medical Center/New York Presbyterian, New York, New York
  - Sorin Medical, P.C., New York, New York

REFERENCES:
- [Result] Lodha A, Giannopoulos S, Sumar R, Ratcliffe J, Gorenchtein M, Green P, Rollefson W, Stout CL, Armstrong EJ. Transradial Endovascular Intervention: Results From the Radial accEss for nAvigation to Your CHosen Lesion for Peripheral Vascular Intervention (REACH PVI) Study. Cardiovasc Revasc Med. 2022 Mar;36:115-120. doi: 10.1016/j.carrev.2021.05.011. Epub 2021 May 15. PMID 34020900

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following physician assessment of patient and general inclusion/exclusion and informed consent signature, subjects were eligible for enrollment pending index procedure inclusion and exclusion criteria.
Groups:
- OAS Use Via Transradial Access (TRA): All patients undergoing peripheral vascular intervention (PVI) via transradial access (TRA) and for whom TRA has been successfully achieved and peripheral lesion deemed appropriate for treatment via TRA per physician discretion.
Period: Overall Study
Arm/Group | OAS Use Via Transradial Access (TRA)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OAS Use Via Transradial Access (TRA)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 10
  White | 33
  Other | 2
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Baseline Rutherford Clinical Category [Count of Participants; unit: Participants]
  Moderate Claudication (2) | 6
  Severe Claudication (3) | 31
  Ischemic Rest Pain (4) | 12
  Minor Tissue Loss (5) | 1

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success:
Description: Successful completion of OA (orbital atherectomy) treatment of target lesion via transradial access without serious transradial access (TRA) related events. Serious TRA related events consist of: Serious TRA site bleeding, serious TRA site hematoma, serious radial artery spasm, serious hand ischemia, stroke, Transient Ischemic Attach (TIA), Serious nerve damage, perforation, TRA site pseudoaneurysm.
Time Frame: Participants were followed from the baseline procedure through the first site-specific standard of care follow-up visit (7-45 days post-procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | OAS Use Via Transradial Access (TRA)
Number analyzed (Participants) | 50
Participants | 49

2. Secondary Outcome: Treatment Success:
Description: Treatment success is defined as <50% residual stenosis post-procedure and without significant angiographic complications without stent placement, or <30% residual stenosis post-procedure and without significant angiographic complications with stent placement.
Time Frame: Participants were followed from baseline procedure through hospital discharge, an expected average of less than 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | OAS Use Via Transradial Access (TRA)
Number analyzed (Participants) | 50
Participants | 49

ADVERSE EVENTS:
Time Frame: The reporting of adverse events (AEs) began immediately after the subject was enrolled through the first standard of care follow-up visit (7 - 45 days post-procedure). For the purposes of this study, pre-planned interventions noted at baseline were not considered reportable AEs.
Description: Adverse events were limited to: SAEs, TRA Related Events, Significant Angiographic Events and OAS and ViperCath device related serious injuries. The reporting of AEs began immediately after the subject was enrolled through study exit.
Arm/Group | OAS Use Via Transradial Access (TRA)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OAS Use Via Transradial Access (TRA) (N=50)
Lower Extremity Disorders (Vascular disorders) | 1 (1) — Peripheral artery restenosis
Procedural Complications, Lower Extremities (Injury, poisoning and procedural complications) | 1 (1) — Peripheral artery restenosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03943160/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03943160/SAP_001.pdf